CLINICAL TRIAL: NCT05618054
Title: Pediatric POTS: Does a Periaqueductal Gray-vagus Nerve Interface Malfunction Explain the Natural History With Its Numerous Co-morbidities?
Brief Title: Periaqueductal Gray-vagus Nerve Interface Malfunction Explain the Natural History With Its Numerous Co-morbidities?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HM20025242
Record Dates: First submitted 2022-11-09; First posted 2022-11-16 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Postural Tachycardia Syndrome
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adolescents with POTS (Other)
  Interventions: Behavioral: Looming task
- Adolescents without POTS (Other)
  Interventions: Behavioral: Looming task

INTERVENTIONS:
Behavioral: Looming task — Participants will be asked to look at some pictures during an fMRI scan. Participants will press a button as soon as they see the image appear.

SUMMARY:
This study is being conducted to see how people with Postural tachycardia syndrome (POTS) make sense of the things they see. The information may help doctors to learn more about how the different parts of people's brains communicate.

ELIGIBILITY:
Inclusion Criteria:

* Females 12-21 years old
* Able to communicate and provide consent/assent
* English speaking
* Diagnosed with POTS (POTS will be defined standardly as a symptomatic ≥ 40 bpm rise in heart rate without a drop in blood pressure and with symptoms of orthostatic intolerance clinically)
* Age-matched healthy control subjects: no POTS or other neurological disorders

Exclusion Criteria:

* Inflammatory arthritis, connective tissue or auto-immune disorder
* Any chronic neurological disorder besides POTS
* Evidence of unstable medical disorder, such as kidney (rising creatinine, or end-stage renal failure) or liver impairment (rising AST or ALT, or end-stage with coagulopathy), poorly controlled significant cardiovascular (CHF), respiratory, endocrine (diabetes - A1c > 9 - or untreated thyroid dysfunction) or uncontrolled psychiatric illness (such as untreated depression, psychosis, etc.)
* Neuropathy, central nervous system disorder (e.g., Cerebral palsy, developmental delay, seizure disorder, MS, stroke, etc.)
* Treatment with a drug or medical device within the previous 30 days that has not received regulatory approval
* Use of hormones (except insulin, thyroid replacement or oral contraceptives, which will be carefully documented)
* Current substance or alcohol abuse
* Any major surgical intervention with general anesthesia in the last 60 days and minor procedure, such as tooth extraction, endoscopy, etc., with local or conscious sedation within 7 days
* Any on-going or pending medical, health or disability related litigation, or current pursuit of disability
* Any condition that in the judgment of the investigator would interfere with the patient's ability to provide informed consent, comply with study instructions, place the patient at increased risk, or which would clearly confound the interpretation of the study results (specific reason will be documented)
* Chronic use of narcotics for pain
* Claustrophobia or any metal hardware that may interfere with MRI
* Investigators and study staff

Ages: 12 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-03-06 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Periaqueductal gray region activation - looming task | 90 minutes
  Functional magnetic resonance imaging (fMRI) will be performed to measure activation of the periaqueductal gray region during the looming task
Periaqueductal gray region activation - resting | 90 minutes
  Functional magnetic resonance imaging (fMRI) will be performed to measure activation of the periaqueductal gray region while at rest

CONTACTS AND LOCATIONS:
Overall Officials: Gisela Chelimsky, M.D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No